CLINICAL TRIAL: NCT02626780
Title: Adipose-derived Stromal Vascular Fraction (SVF) Injections to Stimulate Hair Regrowth for Androgenetic Alopecia
Brief Title: Adipose-derived SVF for Treatment of Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GID BIO, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIDAA-01
Record Dates: First submitted 2015-12-02; First posted 2015-12-10 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SVF Injection (Experimental): Liposuction of a small amount of adipose tissue will be taken from each subject. Stromal Vascular Fraction (SVF) will be disassociated within the GID SVF-2 from the autologous adipose tissue to be injected into a small (approximately 2x2cm) area of the scalp in men or women with androgenic alopecia.
  Interventions: Device: GID SVF-2

INTERVENTIONS:
Device: GID SVF-2 — Comparison of the number of hairs before and after treatment of autologous adipose-derived SVF as a percentage increase or decrease in growth.

SUMMARY:
The general objective of this study is to conduct a safety and feasibility study of a single injection of autologous adipose-derived SVF for the treatment of alopecia.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 - 60 years of age and older that have been diagnosed with androgenetic alopecia.
2. Subjects will be in good health (ASA Class I-II) with a BMI < 35. Must have at least a 2cm x 2cm spot on the scalp which shows evidence of alopecia without scarring or traumatic injury
3. Able and willing to make the required study visits.
4. Able and willing to give consent and follow study instructions.
5. Must speak, read and understand English

Exclusion Criteria:

1. History of bleeding disorders, anticoagulation therapy that cannot be stopped 14 days prior to injection
2. Allergic to lidocaine, epinephrine, valium or sodium phosphate
3. Individuals with a propensity for keloids
4. Individuals with diminished decision-making capacity will not be included in this research study
5. Current use of anti-inflammatory or anticoagulation medications that affect bleeding or are for bleeding disorders. These include: Plavix, Warfarin (Coumadin, Jantoven, Marfarin). In addition, if any of the following medicines are used two (2) weeks prior to surgery the patient will be ineligible.
6. Use of concomitant treatments, including topical medications, oral medications, meso-therapy, non-ablative fractional laser treatment, low-level laser therapy, interfollicular PRP injection and hair transplantation within the preceding 6 months.
7. All smokers and other tobacco users.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-01-22 (Actual); Study Completion 2017-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Maxwell Aesthetics, Nashville, Tennessee
  - Renew Associates, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- SVF Injection: Autologous adipose-derived SVF will be injected into a small (approximately 2x2cm) area of the scalp in men or women with androgenic alopecia.
  GID SVF-2: Comparison of the number and thickness of hair before and after treatment of autologous adipose-derived SVF.
Period: Overall Study
Arm/Group | SVF Injection
Started | 7
Withdrew From Study | 3
Completed | 4
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | SVF Injection
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 41 [21 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
Ludwig Classification Type I [Count of Participants; unit: Participants] — The Ludwig Scale uses 3 different classifications, or Types, to diagnose the severity of female hair loss.
  Type I. Mild hair loss, the frontal hairline remains relatively unaffected. Hair loss may occur on the top and front of the scalp.
  Type II. Moderate hair loss. Thinning, shedding, general decrease in volume, and a center part that continues to widen over time.
  Type III. Extreme hair loss. The scalp is visible to the naked eye.
  Participants | 2
Norwood Classification Type III [Count of Participants; unit: Participants] — Type I. Minimal hair loss.
  Type II. Insignificant hair loss at the temples.
  Type III vertex. Receding hairline and thinning hair on the vertex.
  Type IV. Bigger pattern on the vertex and hairline.
  Type V. Patterns at both sites are bigger but a thin division line is still present.
  Type VI. The bridge is gone but several strands of short fine hair may remain.
  Type VII. The most severe form of hair loss. Little hair on the front or top of the head.
  Participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (Safety)
Description: Subjects will be monitored for Adverse events for the duration of the study.
Time Frame: 6 months
Population: All participants were monitored for adverse events
Measure: Number; unit: adverse events
Arm/Group | SVF Injection
Number analyzed (Participants) | 7
adverse events | 0

2. Secondary Outcome: Growth of New Hair
Description: The change in hair density (number of hairs per square centimeter) from baseline to 6 months after treatment will be expressed as a percentage.
Time Frame: 6 months
Population: Participants that completed 6 month follow-up
Measure: Mean (Standard Deviation); unit: Percentage of hairs/cm^2
Arm/Group | SVF Injection
Number analyzed (Participants) | 4
Percentage of hairs/cm^2 | 31 (9.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SVF Injection
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
This was a small safety and feasibility study, therefore there were no statistical assessments of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT02626780/Prot_SAP_000.pdf